CLINICAL TRIAL: NCT01983540
Title: Evaluation of Antibody Persistence at 3.5 and 4.5 Years of Age in Healthy Children After Primary Series and Booster Vaccination With Investigational (DTaP-IPV-Hep B-PRP~T) or Infanrix Hexa™ Vaccines in Latin America
Brief Title: Antibody Persistence at Age 3.5 and 4.5 Years After Primary and Booster DTaP-IPV-Hep B-PRP~T or Infanrix Hexa Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L28; U1111-1122-2457 (Other: WHO)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type b
Keywords: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Pediatric combined vaccine
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; RIX4414 vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study Group 1 (Experimental): Participants who received 3 doses of DTaP-IPV-Hep B-PRP~T vaccine at 2, 4, 6 months of age concomitantly with Prevenar (PCV7) and Rotarix (2 doses at 2 and 4 months of age), and a booster of the same investigational vaccine concomitantly with Prevenar (PCV7) at 12 to 24 months of age in a previous study.
  Interventions: Biological: DTaP-IPV-Hep B- PRP~T + Prevenar + Rotarix vaccine
- Study Group 2 (Experimental): Participants who received 3 doses of DTaP-IPV-Hep B-PRP~T vaccine at 2, 4, 6 months of age concomitantly with Prevenar (PCV7) and Rotarix (2 doses at 2 and 4 months of age), and a booster of Infanrix hexa vaccine concomitantly with Prevenar (PCV7) at 12 to 24 months of age in a previous study.
  Interventions: Biological: DTaP- IPV-Hep B-PRP~T + Prevenar + Rotarix + Infanrix hexa vaccine
- Study Group 3 (Active Comparator): Participants who received 3 doses of Infanrix hexa vaccine at 2, 4, 6 months of age concomitantly with Prevenar (PCV7) and Rotarix (2 doses at 2 and 4 months of age), and a booster of DTaP-IPV-Hep B-PRP~T vaccine concomitantly with Prevenar (PCV7) at 12 to 24 months of age in a previous study.
  Interventions: Biological: Infanrix hexa + Prevenar + Rotarix vaccine

INTERVENTIONS:
Biological: DTaP-IPV-Hep B- PRP~T + Prevenar + Rotarix vaccine — DTaP-IPV-Hep B-PRP~T vaccine at 2, 4, 6 months of age concomitantly with Prevenar and Rotarix (2 doses at 2 and 4 months of age), and a booster of the same investigational vaccine concomitantly with Prevenar (PCV7) at 12 to 24 months of age in a previous study
  Arms: Study Group 1
Biological: DTaP- IPV-Hep B-PRP~T + Prevenar + Rotarix + Infanrix hexa vaccine — DTaP-IPV-Hep B-PRP~T vaccine at 2, 4, 6 months of age concomitantly with Prevenar and Rotarix (2 doses at 2 and 4 months of age) and a booster dose of Infanrix hexa vaccine with Prevnar at 12 to 24 months of age in a previous study.
  Arms: Study Group 2
Biological: Infanrix hexa + Prevenar + Rotarix vaccine — Infanrix hexa vaccine at 2, 4, 6 months of age concomitantly with Prevenar and Rotarix (2 doses at 2 and 4 months of age), and a booster dose of DTaP-IPV-Hep B-PRP~T vaccine concomitantly with Prevenar vaccine concomitantly with Prevenar at 12 to 24 months of age in a previous study.
  Arms: Study Group 3

SUMMARY:
This is a follow-up of the primary series vaccination schedule in Study A3L24 (NCT01177722) and booster vaccination in Study A3L27 (NCT01444781).

Study Objective:

* To describe the long-term antibody persistence at 3.5 and 4.5 years of age following a 3-dose primary series vaccination of either DTaP-IPV-Hep B-PRP-T+Prevenar™ (PCV7) +Rotarix™ or Infanrix hexa™+Prevenar™ (PCV7) +Rotarix™ vaccination at 2, 4, 6 months of age and a booster vaccination of DTaP-IPV-Hep B-PRP-T+Prevenar™ (PCV7) or Infanrix hexa™+Prevenar™ (PCV7) at 12 to 24 months of age.

Observational Objectives:

* To describe the long-term antibody persistence by group and by stratification on the age at inclusion of the A3L27 booster study.
* To describe the effect of one additional oral dose of stand alone poliovirus isotypes 1, 2 and 3 vaccine* on the antibody persistence immune response for poliovirus isotypes (4 vs 5 doses of poliovirus administered).

DETAILED DESCRIPTION:
No investigational vaccine will be administered in the study. Subjects who were previously randomized and completed the primary series, Study A3L24 and the booster study A3L27 will be invited to take part in this study.

Any serious adverse events (SAEs) related to the vaccines administered during the preceding trial (A3L27;) and SAEs related to A3L28 study procedures will be collected throughout the trial.

No vaccine will be administered as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 years and a half (42 months ± 60 days) on the day of the first study visit
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative (and by independent witness/es if required by local regulations)
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* Receipt of primary vaccination with 3 doses of investigational vaccines during the primary series trial A3L24 (either DTaP-IPV-Hep B-PRP-T or Infanrix hexa, concomitantly administered with Prevenar [PCV7] and Rotarix) and a booster dose during the trial A3L27 (either DTaP-IPV-Hep B-PRP-T or Infanrix hexa, concomitantly administered with Prevenar [PCV7]).

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial visit) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Incomplete primary and booster immunization at trial A3L24 and A3L27
* Receipt of any vaccine in the 4 weeks preceding the first trial visit or planned receipt of any vaccine in the 4 weeks preceding the second trial visit
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Haemophilus influenzae type b infections with other vaccine(s) after completion of A3L27 study
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 3 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Haemophilus influenzae type b infection(s), confirmed either clinically, serologically, or microbiologically after completion of trial A3L27
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating blood drawn
* Acute or chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.

Ages: 42 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 558 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Summary of antibody persistence (for all valences) before the booster doses of DTaP-IPV-Hep B-PRP~T vaccine and Infanrix hexa™ vaccine | Up to 60 days following enrollment
  Anti-D concentrations, ≥0.01 IU/mL, ≥0.1 IU/mL and ≥1.0 IU/mL: Anti-T antibody concentrations ≥0.01 IU/mL, ≥0.1 IU/mL and ≥ 1.0 IU/mL; Anti-Hep B antibody concentrations ≥10 mIU/mL and ≥100 mIU/mL; Anti-PRP antibody concentrations ≥0.15 µg/mL and ≥1.0 µg/mL; Anti-pertussis toxin antibody and anti-filamentous haemagglutinin (FHA) antibody concentrations Lower Limit of Quantitation (LLOQ), ≥2x LLOQ and ≥4x LLOQ and Anti-poliovirus 1, 2, and 3 antibody titers ≥8 (1/dil)

SECONDARY OUTCOMES:
Summary of antibody persistence (for all valences) before the booster doses of DTaP-IPV-Hep B-PRP~T vaccine and Infanrix hexa™ vaccine | Up to 12 months following enrollment
  Anti-D concentrations, ≥0.01 IU/mL, ≥0.1 IU/mL and ≥1.0 IU/mL: Anti-T antibody concentrations ≥0.01 IU/mL, ≥0.1 IU/mL and ≥1.0 IU/mL; Anti-Hep B antibody concentrations ≥10 mIU/mL and ≥100 mIU/mL; Anti-PRP antibody concentrations ≥0.15 µg/mL and ≥1.0 µg/mL; Anti-pertussis toxin antibody and anti-filamentous haemagglutinin (FHA) Ab concentrations LLOQ, ≥2x LLOQ and ≥4x LLOQ and Anti-poliovirus 1, 2, and 3 antibody titers ≥8 (1/dil)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (2):
- Cali, Colombia
- San José, Costa Rica

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com